CLINICAL TRIAL: NCT04567979
Title: Prospective Determination of COVID-19 Infection Rate in Patients With Solid Tumors and Healthcare Workers of the Chemotherapy and Radiotherapy Unit at the Instituto Nacional de Ciencias Médicas y Nutrición Salvador.
Brief Title: Prospective Determination of COVID-19 Infection Rate in a Chemotherapy Unit in Mexico.
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Instituto Nacional de Medicina Genomica (Other Government)
Responsible Party: Principal Investigator, David Huitzil m, Médico Especialista A, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: HEM-3412-20-20-1
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Cancer; Tumor
Keywords: Covid19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with solid tumors: Patients with solid tumors under chemotherapy and / or radiotherapy treatment at our center.
- Healthcare workers: Healthcare workers at the chemotherapy and radiotherapy unit in our center.

SUMMARY:
Cancer patients are considered vulnerable to COVID-19 infection. During the pandemic, cancer patients may need to continue their regular treatment of chemotherapy and / or radiotherapy and therefore must visit a hospital unit. As such, they may be at risk for SARS-CoV-2 infection by means of close contact to other patients and health care workers. Hospitals may implement policies to identify symptomatic subjects and limit their access to the chemotherapy / radiotherapy unit. However, asymptomatic COVID-19 positive patients may escape these filters and potentially be contagious to other patients and their health-related workers that care for other several patients. Therefore, there is a real risk of an outbreak that affects a particularly fragile patient population. Patients and their doctors need to know what is the risk associated to visiting a chemotherapy unit in order to decide if the risk outweighs the benefits of cancer treatment in their particular case. To date, this risk is unknown. The study will test patients and health care workers for COVID-19 infection during the peak of the pandemic in a chemotherapy unit in Mexico in order to determine this risk.

DETAILED DESCRIPTION:
In this is prospective cohort, patients with solid tumors and healthcare workers of the chemotherapy and radiotherapy unit at our center will be followed with a daily digital survey and optionally with biweekly PCR tests for SARS-CoV-2. People with symptoms and / or with a positive PCR test for SARS-CoV-2 will be notified and recommendations according to clinical state will be emitted.

Hypothesis: COVID-19 infection rate among patients with solid tumors treated with chemotherapy and / or radiotherapy will be less than 5% during the pandemic period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors receiving active oncological treatment (chemotherapy, or radiotherapy or biologic therapy) at our center.
* Age: no limit
* Gender: men and women.
* Health-related worker treating patients with solid tumors at the chemotherapy and radiotherapy unit at our center.
* People who sign an informed consent.

Exclusion Criteria:

* Patients with an hematologic cancer.
* Patients with cancer under surveillance or without active oncological treatment, or receiving treatment in another center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer and solid tumors receiving treatment at the chemotherapy and radiotherapy unit, and health-related workers treating these patients.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection rate in patients with solid tumors. | From June 2020 to September 2020.
  Determination of SARS-CoV-2 infection rate among patients with solid tumors treated with chemotherapy and / or radiotherapy during the pandemic period.

OTHER OUTCOMES:
Integration of a cohort of patients with solid tumors receiving oncological treatment. | 4 months
  Identification of patients with solid tumors receiving chemotherapy and / or radiotherapy in our center during the COVID-19 pandemic to get informed consent.
Daily digital follow-up of new-onset respiratory symptoms in the cohort of patients with solid tumors. | 4 months
  To determine the rate of new-onset respiratory symptoms suggestive of COVID-19 among the cohort of patients with solid tumors through a daily digital survey.
SARS-CoV-2 infection rate in the cohort of patients with solid tumors and respiratory symptoms. | 4 months
  To determine the SARS-CoV-2 infection rate in the cohort of patients with solid tumors and respiratory symptoms through a PCR test for SARS-CoV-2.
SARS-CoV-2 infection rate in asymptomatic patients with solid tumors. | 4 months
  To determine the SARS-CoV-2 infection rate in asymptomatic patients with solid tumors through a biweekly PCR test for SARS-CoV-2.
Determination of clinical features and outcomes of cancer patients infected with SARS-CoV-2 . | 4 months
  Determination of demographics, clinical and outcomes of cancer patients infected with SARS-CoV-2.
Integration of a cohort of healthcare workers. | 4 months
  Identification of healthcare workers that treat patients with solid tumors in the chemotherapy and radiotherapy unit at our center to get informed consent.
Daily digital follow-up of new-onset respiratory symptoms in the cohort of healthcare workers. | 4 months
  To determine the rate of new-onset respiratory symptoms suggestive of COVID-19 between the cohort of healthcare workers through a daily digital survey.
SARS-CoV-2 infection rate in the cohort of health-related workers and respiratory symptoms. | 4 months
  To determine the SARS-CoV-2 infection rate in the cohort of healthcare workers with respiratory symptoms through a PCR test for SARS-CoV-2.
SARS-CoV-2 infection rate in asymptomatic healthcare workers. | 4 months
  To determine the SARS-CoV-2 infection rate in asymptomatic healthcare workers through a biweekly PCR test for SARS-CoV-2.
Determination of past infection rate in asymtomatic people through SARS-CoV-2 IgG antibodies detection. | 4 months
  Determination of past infection rate in both cohorts (patients with solid tumors and health-related workers) through IgG antibodies detection at the beginning and at the end of the trial.
Register of oncological patients with solid tumors diagnosed with COVID-19. | 4 months
  To create a register of oncological patients with solid tumors diagnosed with COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel D Huitzil Meléndez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977
- [Result] Zhang L, Zhu F, Xie L, Wang C, Wang J, Chen R, Jia P, Guan HQ, Peng L, Chen Y, Peng P, Zhang P, Chu Q, Shen Q, Wang Y, Xu SY, Zhao JP, Zhou M. Clinical characteristics of COVID-19-infected cancer patients: a retrospective case study in three hospitals within Wuhan, China. Ann Oncol. 2020 Jul;31(7):894-901. doi: 10.1016/j.annonc.2020.03.296. Epub 2020 Mar 26. PMID 32224151
- [Result] Yu J, Ouyang W, Chua MLK, Xie C. SARS-CoV-2 Transmission in Patients With Cancer at a Tertiary Care Hospital in Wuhan, China. JAMA Oncol. 2020 Jul 1;6(7):1108-1110. doi: 10.1001/jamaoncol.2020.0980. PMID 32211820
- [Result] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Result] Desai A, Sachdeva S, Parekh T, Desai R. COVID-19 and Cancer: Lessons From a Pooled Meta-Analysis. JCO Glob Oncol. 2020 Apr;6:557-559. doi: 10.1200/GO.20.00097. No abstract available. PMID 32250659
- [Result] You B, Ravaud A, Canivet A, Ganem G, Giraud P, Guimbaud R, Kaluzinski L, Krakowski I, Mayeur D, Grellety T, Lotz JP. The official French guidelines to protect patients with cancer against SARS-CoV-2 infection. Lancet Oncol. 2020 May;21(5):619-621. doi: 10.1016/S1470-2045(20)30204-7. Epub 2020 Mar 25. No abstract available. PMID 32220659
- [Result] Sidaway P. COVID-19 and cancer: what we know so far. Nat Rev Clin Oncol. 2020 Jun;17(6):336. doi: 10.1038/s41571-020-0366-2. No abstract available. PMID 32265531
- [Result] Burki TK. Cancer guidelines during the COVID-19 pandemic. Lancet Oncol. 2020 May;21(5):629-630. doi: 10.1016/S1470-2045(20)30217-5. Epub 2020 Apr 2. No abstract available. PMID 32247319
- [Result] Marijnen CAM, Peters FP, Rodel C, Bujko K, Haustermans K, Fokas E, Glynne-Jones R, Valentini V, Spindler KG, Guren MG, Maingon P, Calvo FA, Pares O, Glimelius B, Sebag-Montefiore D. International expert consensus statement regarding radiotherapy treatment options for rectal cancer during the COVID 19 pandemic. Radiother Oncol. 2020 Jul;148:213-215. doi: 10.1016/j.radonc.2020.03.039. Epub 2020 Apr 2. No abstract available. PMID 32342861
- [Result] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Result] Qu J, Wu C, Li X, Zhang G, Jiang Z, Li X, Zhu Q, Liu L. Profile of Immunoglobulin G and IgM Antibodies Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Nov 19;71(16):2255-2258. doi: 10.1093/cid/ciaa489. PMID 32337590
- [Result] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501